CLINICAL TRIAL: NCT00506363
Title: The Effect of Different Onset Times of Treatment With 595-nm Pulsed Dye Laser on Improvement of Surgical Scars: A Double Blind Randomised Clinical Trial
Brief Title: Safety and Efficacy of Different Onset Times of Treatment With Pulsed Dye Laser on Improvement of Surgical Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was terminated on May 2008 after inclusion of 10 patients due to low recruitment and patient compliance.
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Center for research and training in skin diseases and leprosy, Tehran University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 423/2224-B
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Scar
Keywords: scar; surgery; lasers
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): pulsed dye laser and dynamic cooling device on the day of suture removal
  Interventions: Procedure: pulsed dye laser therapy
- B (Active Comparator): pulsed dye laser and dynamic cooling device 2 months after suture removal
  Interventions: Procedure: pulsed dye laser therapy
- C (Sham Comparator): dynamic cooling device
  Interventions: Procedure: pulsed dye laser therapy

INTERVENTIONS:
Procedure: pulsed dye laser therapy — Each scar will be divided into 3 equal parts. One part will be randomly allocated to be treated with pulsed dye laser and dynamic cooling device on the day of suture removal. Another part will be treated with pulsed dye laser and dynamic cooling device 2 months after suture removal. Only dynamic cooling device will be used for remaining part serving as control. Treatment will repeat for 6 sessions at 3 weeks intervals.

SUMMARY:
The appearance of skin after surgery plays an important role in patient's self confidence and life style. In fact, Keloids and hypertrophic scars are abnormal wound responses appearing in predisposed individuals after surgery. Among different kind of lasers, used to improve the appearance of hypertrophic scars and keloids, pulsed dye laser is now being used successfully in treatment of scars. Pulsed dye laser is effective in improving the color, height, texture, and elasticity of scars. Also, treatment with this technique is noninvasive, minimally uncomfortable, and requires no anesthesia. This study will assess the efficacy and safety of different onset times of treatment with pulsed dye laser on improvement of surgical scars.

ELIGIBILITY:
Inclusion Criteria:

* Surgical scar with minimum length of 6 cm

Exclusion Criteria:

* History of light sensitivity or photodermatoses
* History of adverse reactions to laser treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
pigmentation, pliability, width and height of surgical scars | baseline, middle of the study, 1 and 3 months after the last treatment session

SECONDARY OUTCOMES:
1- Clinical appearance of scar 2- Patient's satisfaction (scar erythema, scar thickness and scar induration) - Adverse events | 1 and 3 months after the last treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Firooz, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Center for research and training in skin diseases and leprosy, Tehran, Iran

REFERENCES:
- [Background] Nouri K, Jimenez GP, Harrison-Balestra C, Elgart GW. 585-nm pulsed dye laser in the treatment of surgical scars starting on the suture removal day. Dermatol Surg. 2003 Jan;29(1):65-73; discussion 73. doi: 10.1046/j.1524-4725.2003.29014.x. PMID 12534515
- [Background] Conologue TD, Norwood C. Treatment of surgical scars with the cryogen-cooled 595 nm pulsed dye laser starting on the day of suture removal. Dermatol Surg. 2006 Jan;32(1):13-20. doi: 10.1111/1524-4725.2006.32002. PMID 16393593
- [Background] Paquet P, Hermanns JF, Pierard GE. Effect of the 585 nm flashlamp-pumped pulsed dye laser for the treatment of keloids. Dermatol Surg. 2001 Feb;27(2):171-4. doi: 10.1046/j.1524-4725.2001.00169.x. PMID 11207693
- [Background] Alster TS, Williams CM. Treatment of keloid sternotomy scars with 585 nm flashlamp-pumped pulsed-dye laser. Lancet. 1995 May 13;345(8959):1198-200. doi: 10.1016/s0140-6736(95)91989-9. PMID 7739306
- [Background] Alam M, Pon K, Van Laborde S, Kaminer MS, Arndt KA, Dover JS. Clinical effect of a single pulsed dye laser treatment of fresh surgical scars: randomized controlled trial. Dermatol Surg. 2006 Jan;32(1):21-5. doi: 10.1111/1524-4725.2006.32029. PMID 16393594
- [Background] Manuskiatti W, Wanitphakdeedecha R, Fitzpatrick RE. Effect of pulse width of a 595-nm flashlamp-pumped pulsed dye laser on the treatment response of keloidal and hypertrophic sternotomy scars. Dermatol Surg. 2007 Feb;33(2):152-61. doi: 10.1111/j.1524-4725.2006.33033.x. PMID 17300600
- [Derived] Davari P, Gorouhi F, Hashemi P, Behnia F, Ghassemi A, Nasiri-Kashani M, Firooz A. Pulsed dye laser treatment with different onset times for new surgical scars: a single-blind randomized controlled trial. Lasers Med Sci. 2012 Sep;27(5):1095-8. doi: 10.1007/s10103-011-1044-5. Epub 2012 Jan 8. No abstract available. PMID 22228413